CLINICAL TRIAL: NCT05493943
Title: P.E.M.F. Therapy of Chronic Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PEMF Systems, Inc. (Industry)
Collaborators: VA Long Beach Healthcare System (U.S. Federal Agency); Southern California Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VA Protocol 5.9
Record Dates: First submitted 2022-07-13; First posted 2022-08-09 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Chronic Wounds
Keywords: wounds; chronic
MeSH Terms: conditions — Wounds and Injuries; Bronchiolitis Obliterans Syndrome | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 3 arms, 2 have PEMF devices, 1 Control with sham devices
Who Masked: Participant, Care Provider
Masking Description: Random, at time of enrollment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- PEMF low power (Active Comparator): PEMF therapy using a device with low pulse intensity.
  Interventions: Device: Pulsed ElectroMagnetic Field (PEMF) therapy
- PEMF medium power (Active Comparator): PEMF therapy using a medium pulse intensity.
  Interventions: Device: Pulsed ElectroMagnetic Field (PEMF) therapy
- PEMF Sham control (Sham Comparator): Control arm using a sham PEMF device.
  Interventions: Other: Pulsed ElectroMagnetic (PEMF) therapy

INTERVENTIONS:
Device: Pulsed ElectroMagnetic Field (PEMF) therapy — Application of PEMF using treatment coils in eproximity to the area where treatment is desired.
  Arms: PEMF low power; PEMF medium power
Other: Pulsed ElectroMagnetic (PEMF) therapy — Control arm.
  Arms: PEMF Sham control

SUMMARY:
To measure the effectiveness of pulsed electromagnetic fields (PEMF) as an adjunct wound care therapy.

DETAILED DESCRIPTION:
The goal of the three-arm trial is to employ application of pulsed electromagnetic fields (PEMF) directly over chronic wounds combined with standard of care local wound therapy (SOC). Three different PEMF devices, one a low power system (LP-PEMF), another a high power system (HP-PEMF) and the third a sham device that does not emit energy (S-PEMF) will be employed as adjuncts to standard wound care. The primary hypothesis to be tested is that exposure of wounds to one of the PEMF devices leads to significantly better and faster healing than the sham system.

Research Design:

An investigator initiated, prospective, double blinded parallel three arm treatment study. Subjects are randomized to receive one of the three PEMF devices (LP-PEMF, HP-PEMF or sham device) twice daily for 15 minutes directly over a wound. Initially, 40 subjects from each treatment group will be enrolled for total of 120 subjects at VA Long Beach Healthcare System (VALB) at the interim analysis. Based on the results of that analysis, one of the treatment arms will be eliminated and a follow-up study will continue with the remaining two arms. Additional 60 to 100 subjects are to be enrolled after interim analysis and the study may expand to Greater Los Angeles Medical Center. The study is expected to last 2 years.

Participating eligible subjects will be asked to come to the VALB once a week for 14 weeks and then for 2 or 3 visits over 8 more weeks. The total number of visits including the first visit could be up to 17 visits in 5 months. The study has three phases: Screening phase (2 weeks); Treatment phase (12 weeks); and Follow-up phase (8 weeks). Subjects participation in the study may last up to 22 weeks, but subjects who heal early during the Treatment phase will have a reduced period of participation based on when their wound heals.

Methodology

Inclusion criteria include age ≥21 years; presence of venous leg ulcers (VLU), Diabetic foot ulcers (DFU) or Pressure Ulcers (PU); wound size between 2 and 30 cm2; no exposed joint, tendon or bone, no tunneling or sinus tracts; wound duration ≥ 6 weeks.

Each wound will be reviewed for eligibility by assessing with duplex ultrasound, skin changes, tendon/bone/joint involvement, Ankle brachial Pressure Index (ABI), BMI, Hemoglobin A1c, Albumin and other medical history.

Female subjects who are currently breast feeding or capable of conceiving and all males capable of insemination must use an acceptable form of contraception in order to participate in the study (acceptable forms of contraception include condoms for males and contraceptive pills or IUDs for women).

Findings: None

Clinical Significance: Potentially beneficial treatment option for veterans with diabetic foot ulcer, venous leg ulcers or pressure ulcers.

ELIGIBILITY:
Inclusion Criteria

* Age must be at least 21 years old at the time of signing consent. 8.2 The index study ulcer size must be between 2.0 and 30.0 cm2 at the time of randomization. Measurements and photographs will to be taken after sharp debridement if performed at the Randomization Visit.
* The index ulcer must have been present for at least 6 weeks prior to randomization.
* If more than one ulcer is present on the target limb, the largest eligible ulcer should be deemed the study ulcer. Other ulcers close to the study ulcer are allowed and may be of any size. However, they should be > 2cm away from the study ulcer. Ulcers are allowed at other locations such as the on the contralateral limb. Other ulcers present besides the index study wound can be treated with different local care but cannot be treated with the PEMF device.
* Only one site of application of the PEMF device is allowed and the PEMF device must be placed directly over the study ulcer.
* Subjects to be enrolled into the VLU group must have had a duplex ultrasound study (if not done within six months prior the first screening visit) to document venous disease (deep system obstruction or reflux > 0.5 sec, or superficial system reflux > 0.5 sec, or have the characteristic hyperpigmentation and skin changes (lipodermatosclerosis) typical of venous disease.
* Diabetic Foot Ulcer (DFU): Subjects should have with neuropathy demonstrated by monofilament testing and have Wagner grade 1 wounds without involvement of tendon, bone, or joint.
* Pressure Ulcer (PU): PU subject wounds must be stage 3 without deep structure involvement such as bone, tendon, or joint.

Exclusion Criteria

* Wounds due to autoimmune disease such as rheumatoid arthritis or vasculitis.
* Exposed structures deep to the adipose layer of skin such as muscle, fascia, tendon, joint, or bone.
* The presence of sinus tracts that have not been sufficiently marsupialized such that the wound depth cannot be assessed by gross visual inspection is an exclusion.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to complete healing | 12 weeks
  Complete re-epithelization of wound
Wound closure | 12 weeks
  Squared milimeters of wound closure

SECONDARY OUTCOMES:
Number and type of adverse events | 12 weeks
  Safety Endpoint
Device effectiveness | 12 weeks
  Compare the rate of effectiveness between performance of the two PEMF power levels by measuring percentage of wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gordon, MD, PhD, Principal Investigator — VA Long Beach Healthcare System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez MI, Watson PJ, Rowbotham DJ. Effect of pulsed magnetic field therapy on pain reported by human volunteers in a laboratory model of acute pain. Br J Anaesth. 2007 Aug;99(2):266-9. doi: 10.1093/bja/aem129. Epub 2007 May 22. PMID 17519258
- [Background] Salzberg CA, Cooper-Vastola SA, Perez F, Viehbeck MG, Byrne DW. The effects of non-thermal pulsed electromagnetic energy on wound healing of pressure ulcers in spinal cord-injured patients: a randomized, double-blind study. Ostomy Wound Manage. 1995 Apr;41(3):42-4, 46, 48 passim. PMID 7546114
- [Background] Sarma GR, Subrahmanyam S, Deenabandhu A, Babu CR, Madhivathanan S, Kesavaraj N. Exposure to pulsed magnetic fields in the treatment of plantar ulcers in leprosy patients--a pilot, randomized, double-blind, controlled clinical trial. Indian J Lepr. 1997 Jul-Sep;69(3):241-50. PMID 9394172
- [Background] Bragin DE, Statom GL, Hagberg S, Nemoto EM. Increases in microvascular perfusion and tissue oxygenation via pulsed electromagnetic fields in the healthy rat brain. J Neurosurg. 2015 May;122(5):1239-47. doi: 10.3171/2014.8.JNS132083. Epub 2014 Oct 24. PMID 25343187
- [Background] Cheing GL, Li X, Huang L, Kwan RL, Cheung KK. Pulsed electromagnetic fields (PEMF) promote early wound healing and myofibroblast proliferation in diabetic rats. Bioelectromagnetics. 2014 Apr;35(3):161-9. doi: 10.1002/bem.21832. Epub 2014 Jan 3. PMID 24395219
- [Background] Hannemann PF, Mommers EH, Schots JP, Brink PR, Poeze M. The effects of low-intensity pulsed ultrasound and pulsed electromagnetic fields bone growth stimulation in acute fractures: a systematic review and meta-analysis of randomized controlled trials. Arch Orthop Trauma Surg. 2014 Aug;134(8):1093-106. doi: 10.1007/s00402-014-2014-8. Epub 2014 Jun 4. PMID 24895156
- [Background] Matic M, Lazetic B, Poljacki M, Djuran V, Matic A, Gajinov Z. Influence of different types of electromagnetic fields on skin reparatory processes in experimental animals. Lasers Med Sci. 2009 May;24(3):321-7. doi: 10.1007/s10103-008-0564-0. Epub 2008 Jun 7. PMID 18536960
- [Background] Stiller MJ, Pak GH, Shupack JL, Thaler S, Kenny C, Jondreau L. A portable pulsed electromagnetic field (PEMF) device to enhance healing of recalcitrant venous ulcers: a double-blind, placebo-controlled clinical trial. Br J Dermatol. 1992 Aug;127(2):147-54. doi: 10.1111/j.1365-2133.1992.tb08047.x. PMID 1390143
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17519258/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/7546114/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9394172/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25343187/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24395219/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24895156/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18536960/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/1390143/